CLINICAL TRIAL: NCT06185894
Title: Single-step Placenta Accreta Resective Technique Tourniqueted vs Absence, Conservative Uterine Surgery (SPARTACUS) Study
Brief Title: Single-step Placenta Accreta Resective Technique Tourniqueted vs Absence, Conservative Uterine Surgery
Acronym: SPARTACUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdalla Mousa, Lecturer of obgyn Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ms-105-2023
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conservation without the use of a tourniquet (Placebo Comparator): surgical conservation of placenta accreta spectrum cases with Kasr alainy conservative management technique, without the use of a tourniquet
  Interventions: Procedure: Conventional conservative surgery
- conservation with the use of a tourniquet (Active Comparator): surgical conservation of placenta accreta spectrum cases with Kasr alainy conservative management technique, with the use of a uterovesical tourniquet before fetal extraction
  Interventions: Procedure: Uterovesical tourniquet before uterine devascularization steps

INTERVENTIONS:
Procedure: Uterovesical tourniquet before uterine devascularization steps — Insertion of a Foley catheter tourniquet through broad ligament apertures & tightening it immediately before hysterotomy in cases of conservative management of placenta accreta spectrum
  Other Names: Uterine Pringles maneuver
  Arms: conservation with the use of a tourniquet
Procedure: Conventional conservative surgery — Conventional conservative surgery
  Arms: conservation without the use of a tourniquet

SUMMARY:
Background: An optimal international standard for PAS surgery is not yet available, and the establishment of a suitable surgical method is an important focus of in PAS management.

Objective: To assess the efficacy and safety of tourniquet uses for conservative approach in the management of placenta accerta spectrum.

Patients and Methods: 40 pregnant women who underwent conservative management of placenta accrete at Kasr El-Aini hospital (Obstetrics and gynecology department - Faculty of medicine - Cairo university) were included and were divided according to the use of tourniquet into 2 equal groups: Study group (tourniquet group): consists of 20 women for whom tourniquet was used in the lower part of the uterus during surgical treatment of placenta accreta spectrum.Control group (no tourniquet group): consists of 20 women for whom no tourniquet was used.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females with previous CS deliveries (at least 1).
* Patients with ultrasound criteria of placenta accerta spectrum.
* Patients desiring fertility (uterine conservation).
* Patients with gestational age that completed 34 weeks (or more) confirmed by the 1st day of the LMP or 1st trimester ultrasound scan.

Exclusion Criteria:

* Maternal age above 40 years.
* Chronic medical disorders (e.g., cardiac, renal, DM and hepatic diseases).
* Patients presented with severe antepartum hemorrhage (unstable vital signs).
* Patients requested radical management (caesarean hysterectomy).

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Intraoperative quantified blood loss | during operation
  Quantified blood loss estimate with the tourniquet

SECONDARY OUTCOMES:
amount of blood and blood product transfusion | during operation and 48 hours post operative
  amount of blood and blood product transfusion

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

REFERENCES:
- [Derived] Mousa A, Gaafar HM, Abdullah M, Elsherbini MM, Abdel-Rasheed M, Rida D, Saysaneh A, Collins SL, Abdelbar A. Uterovesical tourniquet for conservative management of placenta accreta spectrum: a prospective cohort study in a low-resource setting. BMC Pregnancy Childbirth. 2025 Dec 12. doi: 10.1186/s12884-025-08381-7. Online ahead of print. PMID 41387818